CLINICAL TRIAL: NCT01498913
Title: NovoNorm Post Marketing Surveillance Study
Brief Title: Observational Study of NovoNorm® in Subjects With Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: AGEE-1882
Record Dates: First submitted 2011-12-21; First posted 2011-12-26 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Repaglinide
  Interventions: Drug: repaglinide

INTERVENTIONS:
Drug: repaglinide — Prescription with NovoNorm® 0.5mg, 1mg or 2mg tablets according to product labelling in daily clinical practice at the discretion of the physician

SUMMARY:
This study is conducted in Asia. The aim of this study is to review the safety and efficacy of Novonorm® (repaglinide) in post-marketing use.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean people with diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 5841 (Actual)
Dates: Start 2001-08-30 (Actual); Primary Completion 2005-03-25 (Actual); Study Completion 2005-03-25 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)
2 hours postprandial blood glucose (2-hr PPBG)
Fasting blood glucose (FBG)
Body weight

SECONDARY OUTCOMES:
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Seoul, South Korea

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com